CLINICAL TRIAL: NCT02931084
Title: Natural Course and Recovery After ACL-injury
Acronym: NACOX
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Joanna Kvist, Professor, Linkoeping University
Other Study IDs: NACOX
Record Dates: First submitted 2016-10-09; First posted 2016-10-12 (Estimated); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood, urine and joint fluid will be collected from approximately 120 patientes rom one site of the study
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ACL injury: Patients with an acute (not more than 6 weeks old) anterior cruciate ligament (ACL) injury
  Interventions: Other: Rehabilitation
- ACL reconstruction: Some of the patients with ACL injury will have reconstruction of the ACL. These will be followed as a new group.
  Interventions: Other: Rehabilitation; Procedure: ACL reconstruction

INTERVENTIONS:
Other: Rehabilitation — In line with current treatment guidelines, patients will undergo rehabilitation for at least the first three months, before a decision regarding ACL reconstruction is taken
Procedure: ACL reconstruction — Approximately half of the patients will have ACL-reconstruction after an initial time of rehabilitation
  Groups: ACL reconstruction

SUMMARY:
The natural course after ACL injury is not well described in the literature. Every year about 7000 people, a majority aged 15-30 years old, injure their anterior cruciate ligament (ACL) in Sweden. About 3500 go through surgical treatment and rehabilitation. Despite the large amount of research on ACL-injuries, there are still many patients who have unsatisfactory outcomes regarding instability, decreased activity level, and quality of life, not being able to return to sport as well as an increased risk for osteoarthritis. The general aim of the study is to evaluate the natural course and recovery after ACL injury. Specific aims:

* To evaluate physical, psychological and contextual factors affecting recovery after anterior cruciate ligament (ACL) injury. Recovery is related both to natural course and to treatment chosen
* To evaluate factors affecting the decision for which treatment to choose (ACL reconstruction and rehabilitation or rehabilitation alone)
* To evaluate factors affecting the decision for return to sports
* To study development of knee osteoarthritis after ACL-injury
* To study epidemiology of acute knee trauma
* To study risk factors for new injuries after ACL-injury These aims will be pursued by consequently and prospectively following patients who sustain a new ACL injury in a multicenter study including approximately 800 patients. Assessment methods will be questionnaires to patients, orthopedic doctors and physical therapists. A sub-cohort of 130 patients will undergo multiple clinical and functional examination as well as MRIs and blood, urine and joint fluid samples.

DETAILED DESCRIPTION:
Study design: A descriptive and prospective prognostic cohort study, with consecutive recruitment of patients during a 12 month period from seven sites in Sweden Start of recruiting participants is October 2016. Most participants will receive a diagnosis from an orthopedic doctor approximately 2-4 weeks after their knee injury, and undergo rehabilitation for at least the first three months, before a decision regarding ACL reconstruction is taken (in line with current treatment guidelines). The patient cohort will be naturally divided into reconstruction plus rehabilitation, and rehabilitation only. Being included in the study will not affect the choice of treatment.

Patients will be asked to participate at their initial contact with healthcare, after their knee injury. The recruitment process will differ slightly between the different sites, based on the clinical routine.

Patients who accept to participate will complete web-based questionnaires distributed via smart phones or e-mail, once a week the first 6 weeks, every second week up to 3rd month, every month up to 1 year and every second month up to 3 years after initial injury. The length of the questionnaires varies from very short (approximately 10 questions that take 2 minutes to fill in) to longer at specific critical time points. Each time the patient has contact with an orthopedic surgeon, the patient, orthopedic doctor and physiotherapist (if the patient has contact with one) will be asked to answer a questionnaire about choice of treatment (surgery or not). In addition, when the patient reports that they are back to sport activity, the patient and the physiotherapist will be asked to answer a questionnaire about the decision to return to sport. Patients who will have ACL reconstruction will be followed up with new baseline from the time of reconstruction.

Patients recruited from Linköping will have expanded follow-up data collection at baseline and 3, 6, 12 and 24 months after injury. At these follow-ups, a clinical examination will be completed by an orthopedic surgeon or physiotherapist, MRI, and blood and urine samples will be collected. A joint fluid sample will be acquired at baseline, and at the time of ACL reconstruction (if the patient has surgical treatment). Radiographs will be done at baseline and 5 years follow up. Patients who have ACL reconstruction will be followed up with new baseline at the time for reconstruction, but without MRI or blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a knee injury (ACL injury)
* Age at time of ACL injury: 15-40 years

Exclusion Criteria:

* ACL injury/ACL reconstruction on the same knee
* Serious knee injuries to the injured knee, ex fracture that require separate treatment
* ACL injury more than 6 weeks ago
* Inability to understand written and spoken Swedish language
* Cognitive impairments
* Other illness/injury that impairs function (e.g. fibromyalgia, rheumatic diseases and other diagnosis that causes chronic pain)

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with ACL-injury from 7 different sites in Sweden
Sampling Method: Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Return to physical activity/ sports | 1 year
  Patients report when they are back to unrestricted physical activity or sports
Knee function, IKDC | 1 year
  The IKDC subjective knee evaluation form is a self-administered questionnaire which contains 18 items divided into 3 subgroups. These subgroups are symptoms, sports and daily activities and the patients current and previous levels of knee function.
Osteoarthritis | 5 years
  Development of osteoarthritis examined with x-rays at 5 years
New injuries | 3 years
  Reported new knee injuries
Factors related to treatment choice | 1 year
  Questionnaires to patients, orthopedic surgeon and physical therapist about the treatment decision

SECONDARY OUTCOMES:
Psychological factors affecting recovery | 2 years
  Include questionnaires about motivation, goals, satisfaction, self efficacy, fear for new injury, readiness for return to sports, expectations
Physical factors affecting recovery, Range of motion | 1 year
  Measured with goniometer
IKDC | 2 years
  The IKDC subjective knee evaluation form is a self-administered questionnaire which contains 18 items divided into 3 subgroups. These subgroups are symptoms, sports and daily activities and the patients current and previous levels of knee function.
Physical factors affecting recovery, gait | 4 weeks
  Qualitativ assessment of gait pattern
Physical factors affecting recovery, muscle strength | 6 months
  Measured with the Biodex dynamometer, peak torque at 60 degrees per second
Physical factors affecting recovery, functional performance | 6 months
  Measured with hop tests, evaluated with the LSI (limb symmetry index)
Physical factors affecting recovery, functional performance | 1 year
  Measured with hop tests, evaluated with the LSI (limb symmetry index)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Kvist, Professor, Principal Investigator — IMH Linkoping University, Sweden
Locations (1):
- Linkoping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonesson S, Kuster RP, Kvist J. Accelerometer-assessed physical activity patterns during the first two years after a non-surgically treated ACL injury. Phys Ther Sport. 2023 Nov;64:123-132. doi: 10.1016/j.ptsp.2023.09.011. Epub 2023 Oct 12. PMID 37864852
- [Derived] Sonesson S, Kvist J. Bilateral changes in knee joint laxity during the first year after non-surgically treated anterior cruciate ligament injury. Phys Ther Sport. 2022 Nov;58:173-181. doi: 10.1016/j.ptsp.2022.10.011. Epub 2022 Oct 26. PMID 36368151
- [Derived] Casula V, Tajik BE, Kvist J, Frobell R, Haapea M, Nieminen MT, Gauffin H, Englund M. Quantitative evaluation of the tibiofemoral joint cartilage by T2 mapping in patients with acute anterior cruciate ligament injury vs contralateral knees: results from the subacute phase using data from the NACOX study cohort. Osteoarthritis Cartilage. 2022 Jul;30(7):987-997. doi: 10.1016/j.joca.2022.02.623. Epub 2022 Apr 11. PMID 35421548
- [Derived] Filbay S, Kvist J. Fear of Reinjury Following Surgical and Nonsurgical Management of Anterior Cruciate Ligament Injury: An Exploratory Analysis of the NACOX Multicenter Longitudinal Cohort Study. Phys Ther. 2022 Feb 1;102(2):pzab273. doi: 10.1093/ptj/pzab273. PMID 34939109
- [Derived] Grevnerts HT, Sonesson S, Gauffin H, Ardern CL, Stalman A, Kvist J. Decision Making for Treatment After ACL Injury From an Orthopaedic Surgeon and Patient Perspective: Results From the NACOX Study. Orthop J Sports Med. 2021 Apr 15;9(4):23259671211005090. doi: 10.1177/23259671211005090. eCollection 2021 Apr. PMID 33948447
- [Derived] Kvist J, Gauffin H, Tigerstrand Grevnerts H, Ardern C, Hagglund M, Stalman A, Frobell R. Natural corollaries and recovery after acute ACL injury: the NACOX cohort study protocol. BMJ Open. 2018 Jun 27;8(6):e020543. doi: 10.1136/bmjopen-2017-020543. PMID 29950463